CLINICAL TRIAL: NCT04716127
Title: Benefit From a Proximity-incentive Strategy Based on Vaginal Self-sampling for Women Who do Not Participate to Cervical Cancer Screening in Aude and Hérault [French Departments]: an Interventional Research to Reduce Social and Territorial Inequalities.
Brief Title: A Proximity-incentive Strategy for Cervical Cancer Screening
Acronym: RIDECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Paul Valérie University Montpellier (Unknown); Regional Center for Cancer Screening (CRCDC) - Region of Occitanie - Department of Herault (Unknown); Regional Center for Cancer Screening (CRCDC) - Region of Occitanie - Department of Aude (Unknown); Association for Breast Cancer Screening - Department of Herault (AMHDCS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-A01534-35; RECHMPL20_0133 (Other: Montpellier University Hospital)
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer; Uterine Cervical Disease; Human Papilloma Virus
Keywords: Direct-To-Consumer Screening and Testing; Vaginal self-sampling; HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women 50 to 65 years with no regular cervical cancer screening (Experimental): Women aged 50 to 65 years with no cervical smear or no gynecological examination for more than three years, attending the mobile unit for breast cancer screening in the Department of Hérault, or the Medical and Social Care Center in the Department of Aude.
  Interventions: Behavioral: Proximity-incentive strategy based on vaginal self-sampling for women 50 to 65 years who do not participate to cervical cancer screening

INTERVENTIONS:
Behavioral: Proximity-incentive strategy based on vaginal self-sampling for women 50 to 65 years who do not participate to cervical cancer screening — * Direct offer of a vaginal self-sampling kit with information to perform at home and send back to the laboratory for HR-HPV testing
  * The psychosocial determinants involved in decision-making process and compliance to cervical cancer screening will be collected from open questionnaires and by semi-directive phone interviews
  * Control ; Receive reminder to send the self-sample to the laboratory : After 3 and 6 months without "return", women receive a remind letter to send the vaginal self-sample to the laboratory. We call "return" the receipt of the vaginal self-sample at the laboratory.
  * Control ; Receive reminder to perform cervical smear in case of positive HR-HPV test : In case of a positive HR-HPV test, women are asked to perform a control cervical smear. After 3, 6 months and 12 months without "return", women and their health-care professional will receive a remind letter or a call to perform a cervical smear for control. We call "return" the performance of a pap smear.

SUMMARY:
In France, cervical cancer screening is based on a cervical smear for women aged 25 to 30 years and on High Risk- HPV (HR-HPV) testing for women aged 30 to 65 years. One of the main concerns in France is poor attendance to this screening program, up to 40% of women, which led French Health Authorities to implement population-based organized cervical cancer screening (DO CCU), based on remind letters, starting in 2019.

Our project is a complementary strategy to DO CCU based on direct proposal of a vaginal self-sample device for HR-HPV testing to non-attendee women while attending health care centers. Our hypothesis is that contacting under-screened women directly and proposing them a self-sample device to be used at home will increase their participation to cervical cancer screening.

This project will be held in the Departments of Hérault and Aude, which are among those in the region of Occitanie (south of France) with the lowest participation to cervical cancer screening.

Women aged 50 to 65 years with no cervical smear and/or gynecological examination for more than three years, will be recruited in two sites: in a mobile unit for breast cancer screening implemented in the whole Department of Hérault and in a Medical and Social Care located in a particularly deprived area of Aude (Limoux-Quillan). In each site, non attendee-women will be proposed by a trained mid-wife, a vaginal self-sample device to perform at home and send back by mail to the laboratory of the Hospital of Montpellier, which will perform HR-HPV testing. Women with positive HR-HPV DNA test will be asked to perfom a cervical smear and completion of follow-up will be monitored.

The primary objective of this study will be to evaluate attendance of under-screened women to vaginal self-sampling for cervical cancer screening, i.e. the number of women who accepted a self-sample device among women to whom it has been proposed.

A second objective will be to analyse psycho-social factors associated with cervical cancer screening in this population of non-attendee women, i.e. their socio-economic environment and the way women perceive and are implicated in cervical cancer screening. This secondary objective will be based on a specific questionnaire at recruitment and on semi-directive phone interviews in a sub-group of women. The efficacy of this screening strategy (number of women who performed vaginal self sample and sent it to the laboratory, and number of women who completed follow-up in case of a positive HR-HPV test) will also be monitored.

The number of women to be recruited is 660. The total estimated duration of the project is 60 months, including 24 months for women's recruitment.

Expected results from this project are:

* An increase in participation to cervical cancer screening of non-attendee women aged 50 to 65 years in the Departments of Hérault and Aude.
* Women's education about cervical cancer screening through discussion with the midwife during recruitment and information tools developed for the project
* Information of local health staff and community-based associations about cervical cancer screening and the place of HR-HPV testing.
* Identification of psycho-social factors and potential barriers to compliance to cervical cancer screening.
* Identification of organizational and practical difficulties that must be overcome to improve preventive actions towards deprived populations.

DETAILED DESCRIPTION:
Scientific context :

In France, cervical cancer screening is based on a cervical smear every three years for women aged 25 to 30 years, and on a High-Risk HPV (HR-HPV) detection test every five years for women aged 30 to 65 years. One of the main concerns in France is poor attendance to this screening program. Among non-attendee women, older women (> 50 years old) and women of unfavourable socio-economic conditions are the most represented groups. This observation led French Health Authorities to implement population-based organized cervical cancer screening (DO CCU) starting in 2019. The Departments of Hérault and Aude are among those in Occitanie region (south of France) with the lowest participation to cervical cancer screening. In 2017, a group composed of academics, health professionals, the Regional Center for Cancer Screening in Occitanie and the Association for Breast Cancer Screening in Montpellier-Hérault organized a preliminary study based on a self-questionnaire showing high acceptability of vaginal self-sampling by women aged 25 to 65 years, particularly for women older than 50 years.

The aim of this interventional research is to increase women's participation to cervical cancer screening and to identify psycho-social determinants associated with screening observance. For this purpose, the integrative model of change (Attitude Social Influence Self-efficacy Mode - ASE model) from Vries et al. (2013) seems an interesting model to better understand behavioural changes regarding participation to cervical cancer screening using the proposed strategy.

Research hypothesis:

The project is a proximity-incentive strategy complementary to DO CCU based on direct proposal by a trained mid-wife of a vaginal self-sample device for HR-HPV testing to non-attendee women while attending health care centers. Our hypothesis is that contacting under-screened women directly and proposing them a self-sample device to be used at home along with information on cervical cancer, will increase their participation to cervical cancer screening. Secondary hypotheses are that 1) motivational determinants of ASE and contextual opportunities are associated with the realization of vaginal self-sampling 2) and that vaginal self-sampling is an efficient strategy for cervical cancer screening (i.e. number of self-sampling performed and sent to the laboratory, and number of follow-up for women with a positive HR-HPV DNA test among women who accepted the self-sample device).

Intervention description:

Women aged 50 to 65 years with no cervical smear or no gynecological examination for more than three years will be recruited in two sites: in a mobile unit for breast cancer screening implemented in the whole Department of Hérault and in a Medical and Social Care Center and surrounding areas, located in a particularly deprived area of Aude (Limoux-Quillan). Non attendee-women will be proposed a vaginal self-sample device (Evalyn® brush) to perform at home and send back by mail to the laboratory of the Hospital of Montpellier, which will perform HR-HPV testing using the Cobas 4800 HPV DNA detection test. Women with positive HR-HPV DNA test will be asked to perfom a cervical smear and completion of follow-up will be monitored.

During recruitment, women will complete a questionnaire with the help of a midwife on their socio-economic environment, motivational determinants and on their willingness to perform the vaginal self-sample. These data will be analyzed according to their participation to the proposed screening strategy. In addition, semi-directive interviews will be conducted in a sub-group of women (45 women for each site) to identify the barriers and levers of screening participation.

The number of women to be recruited (i.e. non-attendee women aged 50 to 65 years, who accepted the vaginal self-sample device among those to whom it has been proposed) is 660.

The total estimated duration of the project is 60 months, based on 12 months for preparation of the questionnaires, study subject approvals package and staff recruitment and training, 24 months for women's recruitment, 12 months for follow-up of women with positive HR-HPV DNA test, and data analysis and final report.

Expected Health public impact are (a) an increase in participation to cervical cancer screening of women aged 50 to 65 years in the Departments of Hérault and Aude (b) the development of a proximity-incentive strategy to increase cervical cancer screening within vulnerable populations and populations with limited access to health care in those Departments (c) the identification of psycho social determinants involved in cervical cancer screening attendance (i.e. motivational factors, self-efficacy) (d) the construction of a regional network of professionals involved in cervical cancer screening, including health professionals, field teams, committee-based associations and researchers (e) the development of hypotheses and models for future transferability of this intervention to other Departments of the Occitanie Region as a complement of the national DO CCU program.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic women 50 to 65 years old (50 and 65 years included)
* With no cervical smear (or gynecologic examination) or HPV test for at least 3 years (≥ 3 years)
* Able to understand the study and provide voluntarily a written consent to participate
* Able to understand and answer the questions of the study questionnaire by themselves or with the help of a self-chosen third party
* Beneficiary of social security insurance

Exclusion Criteria:

* Women deprived of their liberty, protected adults or vulnerable persons
* Known cervical lesion or known HPV status
* History of hysterectomy
* History of cervix pathology (conization, laser treatment of the cervix)
* History of cervical cancer
* Known immune-depression

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Attendance of under-screened women to vaginal self-sampling when the self-device is proposed directly | During recruitment
  Number of women who accepted a self-sample device among women to whom it has been proposed

SECONDARY OUTCOMES:
Psychosocial determinants involved in attendance to cervical cancer screening using this screening strategy | During recruitment for the questionnaire and 4 months after recruitment for the semi-directive phone interviews
  The psychosocial determinants (motivation, self-efficacy) involved in decision-making process and compliance to cervical cancer screening will be collected from open questionnaires conducted during women recruitment and later by semi-directive phone interviews for a sub-group of women participating to the study. These data will be organized through a logical model of change.
  The role of socio-economic factors on cervical cancer screening adherence and self-sampling attendance will be evaluated using a validated index of social deprivation (European Deprivation Index - EDI).
Efficacy of the proposed screening strategy | After the last recall letter, sent 6 months after recruitment, if the vaginal self-sample has not been sent to the laboratory
  Number of vaginal self-samples performed and sent to the laboratory for HPV testing by women who accepted the self-sample device
Efficacy of vaginal self-sampling with HPV testing for cervical cancer screening | After the last recall letter, sent 12 months after informing the woman by mail of a positive HR-HPV test, if no cervical smear has been performed
  Number of complete follow-up (cervical smear) obtained among women who had a positive HPV test by vaginal self-sampling

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BOULLE, MD/PhD, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - Arnaud de Villeneuve Hospital, clinical trials Department, Montpellier, Herault
  - Mammobile Hérault, Montpellier

REFERENCES:
- [Derived] Lareyre O, Mollevi C, Broc G, Caspar MN, Pehlivanska G, Boyer H, Groc S, Corradi G, Loy-Morel S, Guy M, Tricheux N, Cousson-Gelie F, Boulle N. An outreach strategy to increase uptake of vaginal self-sampling for cervical cancer screening in older French women: The RIDECA interventional research protocol. Womens Health (Lond). 2024 Jan-Dec;20:17455057241292693. doi: 10.1177/17455057241292693. PMID 39474856